CLINICAL TRIAL: NCT00892684
Title: Omega-3 Fatty Acid Supplementation in Pregnancy and During Lactation: a Randomized, Double-Blind, Placebo Controlled Trial.
Brief Title: Does Omega-3 Fatty Acid Supplementation in Pregnancy and During Lactation Protect the Child From Allergic Disease?
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Linkoeping University (Other Government)
Collaborators: Pharma Nord (Industry); The Ekhaga Foundation, Stockholm, Sweden (Unknown); The Swedish Research Council for Environment, Agricultural Sciences and Spatial Planning (FORMAS) (Other Government); Medical Research Council of Southeast Sweden (Other Government); Ostergotland County Council, Sweden (Other); The Swedish Asthma and Allergy Research Foundation, Stockholm, Sweden. (Unknown)
Responsible Party: Karel Duchén, Linkoeping University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: FA-013
Record Dates: First submitted 2009-05-01; First posted 2009-05-04 (Estimated); Last update posted 2009-05-04 (Estimated); Status verified 2009-05

CONDITIONS: Allergies
Keywords: Randomized; Placebo controlled; Double blind; Omega-3 fatty acids; Pregnancy; Childhood allergy; Cytokines; Eicosanoids; Polyunsaturated fatty acids
MeSH Terms: conditions — Hypersensitivity | interventions — Soybean Oil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Dietary Supplement: Omega-3 long chain polyunsaturated fatty acids — 2.7g ω-3 LCPUFA i.e., 1.6 g EPA and 1.1 g DHA and 23 mg alfa-tocopherol as an antioxidant
  Other Names: Bio-Marin, Pharma Nord, Denmark
Dietary Supplement: Soybean oil (placebo) — 2.8 g soybean oil containing 2.5 g linoleic acid and 0.28 g α-linolenic and 36 mg alfa-tocopherol
  Other Names: Placebo, Pharma Nord, Denmark

SUMMARY:
The incidence of allergic diseases has increased and a relation between allergy and dietary fatty acids has been proposed. Modulation of the maternal immune function during pregnancy may have an impact on future clinical outcomes in the child. The aim of this study was to determine the effects of omega (ω) - 3 long-chain polyunsaturated fatty acid (LCPUFA) supplementation during pregnancy and lactation on the development of allergic disease (i.e., allergic eczema) in the child at 2 years of age. Pregnant women with allergic disease in their immediate family were supplemented daily with 2.7 g ω-3 LCPUFA (n=70) or 2.8 g soybean-oil as placebo (n=75) from gestational week (gw) 25 until the third month of breastfeeding. Skin prick tests, detection of circulating specific IgE antibodies and clinical examinations of the infants were performed at 3, 6, 12 and 24 months of age. The mothers and children were monitored regarding immune modulatory effects during the entire study period.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant woman, at 25 weeks of gestation, with allergic symptoms (rhinitis, conjunctivitis, eczema, asthma or food allergy) herself or the father to be or an older sibling

Exclusion Criteria:

* Soy allergy
* Fish allergy
* Treatment with anti-coagulation
* Commercial omega-3 supplementation

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 146 (Actual)
Dates: Start 2003-03; Primary Completion 2005-06 (Actual); Study Completion 2011-09 (Estimated)

PRIMARY OUTCOMES:
allergic eczema | 2 years

SECONDARY OUTCOMES:
changes in laboratory parameters such as prostaglandins and cytokines associated to the intervention and the primary outcome | 25th gestational week, at partus and 12 months after partus for the mothers, in cord blood at 3, 12 and 24 months for the children

CONTACTS AND LOCATIONS:
Overall Officials: Karel M Duchén, MD, PhD, Principal Investigator — Linkoeping University
Locations (1):
- University Hospital, Linköping, Sweden